CLINICAL TRIAL: NCT03782948
Title: Effect of Robotised Gait Training on Dynamic Balance, Symmetry and Push-off in Persons After Stroke
Acronym: BART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: URIS201802
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: gait training; dynamic balance; gait symmetry; rehabilitation robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (Active Comparator): In each session, the group will undergo standard gait training on BART without pelvic perturbations, i.e.,
  * walk a virtual track on the BART without pelvic perturbations (i.e., the pelvic brace of the BART device will be set to follow the patient's motion) for 10 minutes;
  * practise gait symmetry and take-off using visual feedback without pelvic perturbations in two 10-minute sessions.
  Interventions: Device: Standard gait training on BART without pelvic perturbations
- Experimental (Experimental): In each session, the group will undergo robotised gait training with BART with pelvic perturbations, i.e.,
  * walk a virtual track on the BART with pelvic perturbations during virtual uphill walk and virtual curved walk for 10 minutes;
  * practise gait symmetry and take-off using visual feedback with pelvic perturbations for 10 minutes;
  * practise dynamic gait balance using pelvic perturbations during treadmill walking for 10 minutes.
  Interventions: Device: Robotised gait training with BART with pelvic perturbations

INTERVENTIONS:
Device: Standard gait training on BART without pelvic perturbations — The Balance Assisted Robot on Treadmill (BART) enables various types of gait training on treadmill with visual feedback. It interfaces to the pelvis of the walking subject in an actuated and admittance-controlled manner, thus providing transparent haptic interaction with negligible power transfer.
  Arms: Controls
Device: Robotised gait training with BART with pelvic perturbations — In addition to the standard gait training, the BART will deliver perturbations in the forward/backward and left/right direction.
  Arms: Experimental

SUMMARY:
Rehabilitation robotics is increasingly used because it enables the patients to practice a wide array of movements. Dynamic balance training is essential for gait rehabilitation and robotised devices enhance repeatability, objectivity and precision of such training combined with monitoring and recording of kinematic and kinetic data. The aim of the study is to explore the effect of robot-assisted gait training on dynamic balance, symmetry and take-off in patients after stroke. The investigators will conduct a randomised intervention study where one group will receive visual feedback on gait status and the other group will receive kinetically-assisted training using a robotised device in addition to the visual feedback.

DETAILED DESCRIPTION:
Gait training will start 3 weeks after admission to inpatient rehabilitation. It will last for 3 weeks, 5 times per week, 30 minutes per day. The first few sessions with the robotic device will serve to familiarise the patient with the BART device and training conditions. Further details are described in the Arms and Interventions section.

ELIGIBILITY:
Inclusion Criteria:

* Subacute phase after first ischaemic or haemorrhagic stroke (less than 6 months after stroke);
* Limb hemiparesis;
* Ability to walk independently (FAC 6) or with assistance (FAC 5) on flat and uneven surfaces, stairs and slopes;
* Adequate cardiovascular ability (NYHA 1).

Exclusion Criteria:

* Degenerative process or postoperative condition on lower-limb joints that would hinder gait;
* Associated neurological disease;
* Decreased cognitive ability (KPSS < 25).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in postural stability during walking | Assessment before and after the 3-week training programme
  Assessed using the Functional Gait Assessment (FGA) scale. The scale scores range from 0 to 30, with higher scores indicating less impairment.

SECONDARY OUTCOMES:
Change in functional ambulation category | Assessment before and after the 3-week training programme
  Assessed using the Functional Ambulation Categories (FAC) scale. The FAC is a 6-point scale (0-5), with higher category indicating better walking ability.
Change in functional independence | Assessment before and after the 3-week training programme
  Assessed using the Motor subscale of the Functional Independence Measure (FIM). FIM Motor subscale scores range from 13 to 91, with higher scores indicating better functional independence.
Change in fall-risk related mobility | Assessment before and after the 3-week training programme
  Assessed using the Timed Up and Go (TUG) test. Longer TUG times indicate worse mobility (and thus higher fall risk).
Change in ability to change directions while stepping | Assessment before and after the 3-week training programme
  Assessed using the Four Square Step Test (FSST). The FSST is timed, with longer times indicating worse ability.
Change in walking speed over a short distance | Assessment before and after the 3-week training programme
  Assessed using the 10 Meter Walk Test (10MWT)
Change in walking speed over a long distance | Assessment before and after the 3-week training programme
  Assessed using the 6 Minute Walk Test (6MWT)

OTHER OUTCOMES:
Changes in kinesiological characteristics of gait | Assessment before and after the 3-week training programme
  Assessed using the BART device

CONTACTS AND LOCATIONS:
Overall Officials: Matjaž Zadravec, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia